CLINICAL TRIAL: NCT03716232
Title: The Safety and Efficacy of a Short Specially Designed Fully Covered Metallic Stent in the Management of Benign Post-surgical Biliary Strictures: a Randomized-controlled Study
Brief Title: Kaffes Stent in the Management of Post-surgical Biliary Strictures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Theodor Bilharz Research Institute (Other); National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Hany Shehab, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPB01
Record Dates: First submitted 2018-10-13; First posted 2018-10-23 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Benign Biliary Stricture; Biliary Stricture; Cholangitis; Bile Duct Stricture; Bile Duct Injury
MeSH Terms: conditions — Cholangitis | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple plastic stents (Active Comparator): * All procedures will be performed under propofol sedation. Strictures will be identified by cholangiography and then dilated by a dilating balloon (diameter 6-10mm). A 10 French plastic stent will be inserted bypassing the level of the stricture.
  * Stent replacement and the addition of further stents will be planned after 3 months from the initial procedure and every 3 months until stricture resolution occurs with a maximum of four procedures. Balloon dilatation with a 6-10 mm balloon will be used in each session before stent insertion.
  Interventions: Device: Multiple plastic stents
- Metallic stent (Experimental): All procedures will be performed under propofol sedation. Strictures will be identified by cholangiography and then dilated by a dilating balloon (diameter 6-10mm). A 4-6cm fully covered expandable metallic stent (Kaffes stent, Taewoong medical, Seoul, Korea) will then be deployed at the level of the stricture. In cases close to the hepatic hilum where the deployment of the stent is expected to reach one duct and possibly block another duct, a 7 Fr stent will be inserted prior to deployment of the metallic stent in the contralateral duct..
  - Stent will be extracted endoscopically after 6 months.
  Interventions: Device: Metallic stent

INTERVENTIONS:
Device: Metallic stent — All procedures will be performed under propofol sedation. Strictures will be identified by cholangiography and then dilated by a dilating balloon (diameter 6-10mm). A 4-6cm fully covered expandable metallic stent (Kaffes stent, Taewoong medical, Seoul, Korea) will then be deployed at the level of the stricture. In cases close to the hepatic hilum where the deployment of the stent is expected to reach one duct and possibly block another duct, a 7 Fr stent will be inserted prior to deployment of the metallic stent in the contralateral duct..
  - Stent will be extracted endoscopically after 6 months.
  Arms: Metallic stent
Device: Multiple plastic stents — Strictures will be identified by cholangiography and then dilated by a dilating balloon (diameter 6-10mm). A 10 French plastic stent will be inserted bypassing the level of the stricture.
  Stent replacement and the addition of further stents will be planned after 3 months from the initial procedure and every 3 months until stricture resolution occurs with a maximum of four procedures. Balloon dilatation with a 6-10 mm balloon will be used in each session before stent insertion.
  Arms: Multiple plastic stents

SUMMARY:
Post-surgical biliary strictures are common especially after cholecystectomy. Standard treatment involves the performance of multiple procedures over a 1 year period at least using several plastic stents to achieve permanent dilatation of these strictures.

Metallic stents have the theoretical benefit of absence of need of multiple sessions.

These strictures however are frequently very close to the hilum and thus previously considered a contraindication for insertion of metallic stents for the fear of occlusion of the contralateral ducts. Metallic stent migration is also a frequent problem.

The use of a metallic stent that is short and completely intraductal, in theory, should reduce the risk of stent migration.

This is a randomized controlled trial comparing the efficacy and safety of a short metallic intraductal stent to the conventional treatment which is multiple plastic stents. In cases with a stricture reaching or close to the hilum a technique is used to avoid obstruction of the contralateral ducts which is insertion of a 7 French plastic stent alongside the metallic stent.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed benign postsurgical biliary stricture by presence of all 3 of the following:

Ultrasound imaging or Magnetic resonance cholangiopancreatography (MRCP) showing biliary dilatation, Raised bilirubin and or alkaline phosphatase, History of biliary tree surgery within the previous year

* Naïve to endoscopic therapy
* Age > 18 years

Exclusion Criteria:

* Coagulopathy
* Inability of patient to adhere to regular follow-up
* Living-donor liver transplant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 6 months after removal of stents
  Proportion of patients with Absence of clinical or laboratory evidence of recurrence of biliary obstruction

SECONDARY OUTCOMES:
Technical success | At time of procedure
  Proportion of patients with Successful deployment of stents
Stricture resolution at end of treatment | After 6 months in the metallic stent group and after 12 or 15 months in the multiple plastic stents group
  Radiological resolution of the stricture at the time of removal of the stents (after insertion of 3 or 4 stents) and after removal of the metallic stent.
Occurrence of complications | up to 6 months after the last procedure
  occurence of any procedure-related complication

CONTACTS AND LOCATIONS:
Overall Officials: hany shehab, FRCP, Principal Investigator — Cairo University
Locations (3):
- Egypt (3):
  - Kasr Alaini University Hospital, Cairo, New Cairo
  - National hepatology and tropical medicine research institute, Cairo
  - Theodor Bilharz Institute, Cairo